CLINICAL TRIAL: NCT03107299
Title: Evaluation of the Impact of 3 Methods of Communication on the Adherence of Methotrexate in Patients With Rheumatoid Arthritis
Acronym: METHO-PR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2016_843_0006
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Methotrexate; Polyarthritis; Rheumatoid
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other)
  Interventions: Other: Communication methods to encourage adherence
- Send sms to patients (Other)
  Interventions: Other: Communication methods to encourage adherence
- pharmaceutical maintenance following medical consultation (Other)
  Interventions: Other: Communication methods to encourage adherence

INTERVENTIONS:
Other: Communication methods to encourage adherence — Prospective randomized controlled study in intention to treat in open monocentric in 3 arms: all patients benefiting from the current management (medical consultation every 4 to 6 months in the department of rheumatology)

SUMMARY:
Methotrexate (MTX) is the first-line treatment for rheumatoid arthritis (RA). Poor adherence of this treatment decreases the control of the disease and the effectiveness of the associated treatments.

The aim would be to study the observance of patients with RA and to be able to propose adequate solutions favoring patient compliance and thus the stability of the pathology.

For this purpose, 3 methods of communication have been put in place to encourage adherence: usual care by the rheumatologist, sms sending or pharmaceutical maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients attending Day Hospital or consultation of rheumatology with rheumatoid polyarteritis and under treatment with MTX alone or in combination with another therapeutic, fixed dosage for at least 3 months.
* Consenting Patient
* Literate French-speaking patient,
* Patient with a mobile phone
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient not managing his own treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
CQR19 (Compliance Questionnaire Rheumatology) Compliance Measurement Surveywith rheumatoid arthritis. | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Derived] Mary A, Boursier A, Desailly Henry I, Grados F, Sejourne A, Salomon S, Fardellone P, Brazier M, Goeb V. Mobile Phone Text Messages and Effect on Treatment Adherence in Patients Taking Methotrexate for Rheumatoid Arthritis: A Randomized Pilot Study. Arthritis Care Res (Hoboken). 2019 Oct;71(10):1344-1352. doi: 10.1002/acr.23750. PMID 30192070